CLINICAL TRIAL: NCT04936984
Title: An Open-Label, Randomized, 4-Period Crossover Study Evaluating the Bioequivalence of Two Abaloparatide-sMTS Treatments and the Effect of Small Variations in Wear-Time in Healthy Women.
Brief Title: Study to Evaluate and Compare the Bioequivalence of Two Abaloparatide-sMTS Treatments in Healthy Women.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radius Health, Inc. (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BA058-05-023
Record Dates: First submitted 2021-06-16; First posted 2021-06-23 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-06

CONDITIONS: Osteoporosis
Keywords: osteoporosis; transdermal delivery; microneedle patch; solid microstructured transdermal system; abaloparatide TYMLOS®; abaloparatide-SC; PK
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Intervention Model Description: All subjects were to receive a transdermal patch containing 300 μg abaloparatide for 4,5 and 7 minutes in 4 separate periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Patheon sMTS 5 min, then by Kindeva sMTS 5 min, then Patheon sMTS 4 min, then Patheon sMTS 7 min (Experimental): Abaloparatide-sMTS is a drug-device combination product consisting of abaloparatide coated onto a microstructure array for transdermal administration of abaloparatide. The abaloparatide-sMTS is manufactured at Patheon (sterile environment) or Kindeva (low bioburden environment).
  Interventions: Combination Product: abaloparatide-sMTS (Patheon); Combination Product: abaloparatide-sMTS (Kindeva)
- Kindeva sMTS 5 min, then Patheon sMTS 7 min, then Patheon sMTS 5 min, then Patheon sMTS 4 min (Experimental): Abaloparatide-sMTS is a drug-device combination product consisting of abaloparatide coated onto a microstructure array for transdermal administration of abaloparatide. The abaloparatide-sMTS is manufactured at Patheon (sterile environment) or Kindeva (low bioburden environment).
  Interventions: Combination Product: abaloparatide-sMTS (Patheon); Combination Product: abaloparatide-sMTS (Kindeva)
- Patheon sMTS 4 min, then Patheon sMTS 5 min, then Patheon sMTS 7 min, then Kindeva sMTS 5 min (Experimental): Abaloparatide-sMTS is a drug-device combination product consisting of abaloparatide coated onto a microstructure array for transdermal administration of abaloparatide. The abaloparatide-sMTS is manufactured at Patheon (sterile environment) or Kindeva (low bioburden environment).
  Interventions: Combination Product: abaloparatide-sMTS (Patheon); Combination Product: abaloparatide-sMTS (Kindeva)
- Patheon sMTS 7 min, then Patheon sMTS 4 min, then Kindeva sMTS 5 min, then Patheon sMTS 5 min (Experimental): Abaloparatide-sMTS is a drug-device combination product consisting of abaloparatide coated onto a microstructure array for transdermal administration of abaloparatide. The abaloparatide-sMTS is manufactured at Patheon (sterile environment) or Kindeva (low bioburden environment).
  Interventions: Combination Product: abaloparatide-sMTS (Patheon); Combination Product: abaloparatide-sMTS (Kindeva)

INTERVENTIONS:
Combination Product: abaloparatide-sMTS (Patheon) — single-dose administration of abaloparatide 300 μg applied to the thigh for 5 minutes
  Other Names: abaloparatide-sMTS
Combination Product: abaloparatide-sMTS (Kindeva) — single-dose administration of abaloparatide 300 μg applied to the thigh for 5 minutes
  Other Names: abaloparatide-sMTS
Combination Product: abaloparatide-sMTS (Patheon) — single-dose administration of abaloparatide 300 μg applied to the thigh for 4 minutes
  Other Names: abaloparatide-sMTS
Combination Product: abaloparatide-sMTS (Patheon) — single-dose administration of abaloparatide 300 μg applied to the thigh for 7 minutes
  Other Names: abaloparatide-sMTS

SUMMARY:
A study to evaluate the bioequivalence of abaloparatide between 2 abaloparatide-sMTS treatments 300 μg treatments applied to the thigh for 5 minutes.

DETAILED DESCRIPTION:
This is a single site, open-label, randomized, 4-period crossover study to evaluate the bioequivalence of 2 abaloparatide-sMTS 300 μg treatments (Patheon sterile abaloparatide-sMTS and Kindeva ultra-low bioburden abaloparatide-sMTS) applied to the thigh for 5 minutes. The study will also evaluate the effect of small deviations in the wear-time of the Patheon abaloparatide-sMTS worn for 4 minutes or 7 minutes compared to the Patheon abaloparatide-sMTS worn for the prescribed 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged 40 to 65 years old, inclusive, at Screening
* Good general health as determined by medical history and physical exam (including vital signs, and has a body mass index between 18 and 34 kg/m^2 inclusive)
* Laboratory tests within the normal range
* Serum 25-hydroxyvitamin D values must be > 20 ng/mL

Exclusion Criteria:

* Presence or history of any disorder that may prevent the successful completion of the study.
* Diagnosed with osteoporosis, Paget's disease, or other metabolic bone diseases (eg, vitamin D deficiency or osteomalacia), or had a non-traumatic fracture within 1 year prior to the initial screening;
* History of any cancer within the past 5 years other than squamous or basal cell carcinoma;
* History of allergy to abaloparatide or drugs in a similar pharmacological class;

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2021-08-13 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | 4 single-dose administrations, separated by 48 hours.
Area under the plasma concentration-time curve (AUC) from time 0 to the time of the last quantifiable concentration (AUC 0-t) | 4 single-dose administrations, separated by 48 hours.
AUC from time 0 extrapolated to time infinity (AUC 0-∞) | 4 single-dose administrations, separated by 48 hours.

SECONDARY OUTCOMES:
Subjects with treatment-emergent AEs and SAEs | 14 ± 2 days

CONTACTS AND LOCATIONS:
Locations (1):
- Medpace Clinical Pharmacology, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No